CLINICAL TRIAL: NCT01818739
Title: Detection of Sentinel Lymph Nodes in Patients With Endometrial Cancer Undergoing Robotic-Assisted Staging: Comparison of Isosulfan Blue and Indocyanine Green Dyes With Fluorescence Imaging
Brief Title: Lymph Node Mapping in Patients With Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Floor Backes, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-12114; NCI-2013-00530 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-14; First posted 2013-03-26 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Robotic-Assisted Staging
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Indocyanine Green; iso-sulfan blue; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- sentinel lymph node detection (Experimental): Patients undergo sentinel lymph node detection using fluorescence imaging with indocyanine green solution and isosulfan blue and sentinel lymph node biopsy.
  Interventions: Procedure: sentinel lymph node detection; Drug: indocyanine green solution; Drug: isosulfan blue; Procedure: sentinel lymph node biopsy

INTERVENTIONS:
Procedure: sentinel lymph node detection — Undergo sentinel lymph node detection using fluorescence imaging with indocyanine green solution and isosulfan blue
Drug: indocyanine green solution — Undergo sentinel lymph node detection using fluorescence imaging with indocyanine green solution and isosulfan blue
  Other Names: IC-GREEN; ICG solution
Drug: isosulfan blue — Undergo sentinel lymph node detection using fluorescence imaging with indocyanine green solution and isosulfan blue
  Other Names: Lymphazurin; N-[4-[4-(diethylamino)phenyl] (2,5-disulfophenyl) Methylene]-2,5-cyclohexadien-1-ylidene]-N-ethylethanaminium hydroxide
Procedure: sentinel lymph node biopsy — Undergo sentinel lymph node biopsy
  Other Names: sentinel node biopsy

SUMMARY:
This clinical trial studies lymph node mapping in patients with endometrial cancer. Lymph node mapping may allow for limited removal of lymph nodes in as part of endometrial cancer staging and treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the negative predictive value of pelvic sentinel lymph node (SLN) in endometrial cancer to predict nodal metastasis.

SECONDARY OBJECTIVE:

II. To examine the ability of sentinel lymph nodes to increase the detection of metastatic disease through ultra-sectioning and immuno-histochemical (IHC) staining by comparing IHC results and standard hematoxylin and eosin (H&E) results.

OUTLINE:

Patients undergo sentinel lymph node detection using fluorescence imaging with indocyanine green solution and isosulfan blue and sentinel lymph node biopsy and detection of sentinel lymph nodes is noted in the within 30 minutes of injection of the dye, followed by full pelvic lymph node dissection and aortic lymph node dissection as indicated, and standard hysterectomy and salpingo-oophorectomy.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years for a total of 5 years according to the standard surveillance guidelines for endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be willing and able to provide informed consent
* The patient is willing and able to comply with the study protocol
* The patient has endometrial cancer and is scheduled for robotic hysterectomy and lymphadenectomy
* The patient agrees to follow-up examinations out to 5-years post-treatment

Exclusion Criteria:

* The patient is not a candidate for robotic assisted hysterectomy and lymphadenectomy
* The patient has known or suspected allergies to iodine, indocyanine green (ICG) or isosulfan blue (ISB)
* The patient has hepatic dysfunction confirmed by bilirubin > 2 x normal (based on reference values from the laboratory used by the patient)

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Floor Backes, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Background] Backes FJ, Cohen D, Salani R, Cohn DE, O'Malley DM, Fanning E, Suarez AA, Fowler JM. Prospective clinical trial of robotic sentinel lymph node assessment with isosulfane blue (ISB) and indocyanine green (ICG) in endometrial cancer and the impact of ultrastaging (NCT01818739). Gynecol Oncol. 2019 Jun;153(3):496-499. doi: 10.1016/j.ygyno.2019.03.252. Epub 2019 Apr 4. PMID 31230614
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened in February 2013 and patients were enrolled between March 2013 and November 2016
Period: Overall Study
Arm/Group | Sentinel Lymph Node Detection
Started | 204
Completed | 204
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients received dye injections
Arm/Group | Sentinel Lymph Node Detection
Number analyzed (Participants) | 204
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 204
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 36.5 [18.2 to 65.6]

OUTCOME MEASURES:

1. Primary Outcome: Negative Predictive Value of Sentinel Lymph Node Prediction of Metastatic Disease
Description: NPV is found by dividing the number of true negatives by the number of all patients without pelvic lymph node metastases. Exact 95% confidence intervals (CIs) for the proportions will be calculated.
Time Frame: average of 1-14 days after the procedure when final pathologic evaluation has been completed
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Sentinel Lymph Node Detection: Patients with negative SLN who underwent sentinel lymph node detection using fluorescence imaging with indocyanine green solution and isosulfan blue and sentinel lymph node biopsy.
Arm/Group | Sentinel Lymph Node Detection
Number analyzed (Participants) | 163
percentage of patients | 98.8 [95.5 to 99.7]

2. Secondary Outcome: Percentage of Metastatic Cases Found Using Ultra-sectioning and IHC Staining
Description: The percentage of metastatic cases analyzed by H&E will be compared to those of H&E-plus- IHC/ultrastaging using a "z-test".
Time Frame: average of 1-14 days after the procedure when final pathologic evalulation has been completed
Measure: Number; unit: percentage of patients with positive LN
Arm/Group | Sentinel Lymph Node Detection
Number analyzed (Participants) | 204
percentage of patients with positive LN | 17

ADVERSE EVENTS:
Arm/Group | Sentinel Lymph Node Detection
All-Cause Mortality (participants affected / at risk) | 0/204
Serious Adverse Events (participants affected / at risk) | 0/204
Other Adverse Events (participants affected / at risk) | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes